CLINICAL TRIAL: NCT01791283
Title: Real-time Comparison of Left Ventricular Strokevolume Measurement by Four Different Methods
Acronym: FourComp
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Anna Oscarsson, MD, PhD, University Hospital, Linkoeping
Other Study IDs: FourCompv1
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Difference in Measured Results Using Four Different Strokevolume Measurements Simultaneously.
Keywords: Left ventricular stroke volume; Arterial waveform analysis; Esofageal doppler; Ultrasound; Cardiac magnetic Imaging; Limits of agreement
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volounteers with no previous medical history, age between 20-40. Both male and female. Subjects are provided extensive information about the study and the obligations and expectations included. All subjects sign a witnessed informed consent before inclusion.
  Interventions: Procedure: Arterial waveform analysis, esofageal doppler, transthoracal cardiac ultrasound, Cardiac magnetic resonance imaging.

INTERVENTIONS:
Procedure: Arterial waveform analysis, esofageal doppler, transthoracal cardiac ultrasound, Cardiac magnetic resonance imaging.
  Other Names: Vigileo/FloTrac, Edward Lifesciences (arterial waveform analysis); CardioQ, Deltex medical (esofageal doppler); Philips, Magnetic Resonance Imaging; Vivid S6, GE, Cardiac ultrasound

SUMMARY:
Real-time comparison of three different bedside strokevolumemeasurements (arterial waveform analysis, eosofageal doppler and 2D transthoracal ultrasound) validated against cardiac magnetic resonance imaging (CMRI)

DETAILED DESCRIPTION:
20 healthy volounteers between age of 20-40 years, no previous medical history undergo simoultaneous left ventrikular strokevolume measurements using three different methods at rest. After datasampling and without moving, the subject then undergo Cardiac Magnetic Resonance Imaging with 2D-throughplane and cine tecnology for validation of volume measurements. The data is then analyzed using Bland-Altman calculation.

ELIGIBILITY:
Inclusion Criteria:Healthy volounteers age 20-40, BMI < 30, weight < 100 kg, no medications, sinus rythm on ECG, no contra-indications for MRI, ability to give written informed consent.

-

Exclusion Criteria:

* Heart and/or vascular disease such as angina pectoris, arrythmias, claudicatio intermittens e g.
* Diseases in gastrointestinal tract or nose.
* Coagulopathies
* Pregnancy
* Allergys for local anaesthetics
* Claustrofobia

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volounteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Limits of agreement (LOA) is less than 30% using CMRI as validation for each individual measurement of left ventricular stroke volume. | Study period (1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Liffner, MD, Principal Investigator — Intensivvardskliniken, Linkoping University Hospital
Locations (1):
- Departement for intensive care medicine, Universitetssjukhuset, Linköping, Sweden